

Study Number: 2022-0938

Page 1 of 22

#### Informed Consent/Authorization for Participation in Research

**Title of Research Study:** A phase 1 study of JV-213 autologous

CD79b-targeting chimeric antigen receptor T-

cell therapy in adults with relapsed or

refractory B-cell lymphomas

**Study Number:** 2022-0938

Principal Investigator: Sattva Neelapu

Participant's Name Medical Record Number

#### **Key Information**

The following is a short summary of this study to help you decide whether or not to be a part of this study. More detailed information is listed later on in this form.

#### Why am I being invited to take part in a research study?

You are invited to take part in a research study because you have B-cell lymphoma that is relapsed (has come back) or refractory (has stopped responding to treatment).

#### What should I know about a research study?

- Someone will explain this research study to you.
- Whether or not you take part is up to you.
- You can choose not to take part.
- You can agree to take part and later change your mind.
- Your decision will not be held against you.
- You can ask all the questions you want before you decide.

#### Why is this research being done?

The goal of this clinical research study is to find the highest tolerable dose of JV-213 (a type of autologous CAR T cell therapy) that can be given to patients who have B-cell lymphoma that is relapsed or refractory. The safety and possible effects of JV-213 will also be studied.



JV-213 is made from your T cells (a type of white blood cell) which are collected from you and then genetically modified (changed) in a lab to help better recognize the cancer cells in your body and attack them.

This is the first study of JV-213 in humans.

This is an investigational study. JV-213 is not FDA approved or commercially available. It is currently being used for research purposes only. It is considered investigational to give JV-213 to treat B-cell lymphomas that have either come back or gotten worse after other treatments. As part of this study, you will also receive conditioning chemotherapy (fludarabine and cyclophosphamide) to help prepare your body to receive JV-213. Both fludarabine and cyclophosphamide are FDA approved and commercially available for this purpose.

The study doctor can explain how the study drugs are designed to work in more detail.

#### How long will the research last and what will I need to do?

Your participation in this study may last up to about 15 years, depending on how you respond to the study drug. During the study, you may be hospitalized for about 7 days. After being released from the hospital, you will be expected to come to the clinic about 12 times over the first 2 years and every year after that for up to 15. Follow-ups after the 5<sup>th</sup> year may be done as an in-person clinic visit or by video/telephone encounter or by mailed questionnaire.

You will be asked to have physical exams, blood tests, imaging scans, tumor and/or bone marrow biopsies, and a leukapheresis procedure as part of the study.

More detailed information about the study procedures can be found under "What happens if I agree to be in this research?"

#### Is there any way being in this study could be bad for me?

Before choosing to take part in this study, you should talk to the study team about your concerns, including side effects, additional tests/procedures (such as biopsies or blood draws) outside of your normal medical care, potential expenses, hospitalization, and time commitment.

More detailed information about the risks of this study can be found under "Is there any way being in this study could be bad for me? (Detailed Risks)"

Will being in this study help me in any way?



The study drug may help to control the disease. Future patients may benefit from what is learned. However, it cannot be promised that there will be any benefits to you or others from your taking part in this research.

#### What happens if I do not want to be in this research?

Participation in research is completely voluntary. You can decide to participate, not participate, or discontinue participation at any time without penalty or loss of your regular benefits.

Instead of taking part in the study, you may choose to receive chemotherapy, radiation therapy, or other drug therapy, including FDA-approved CAR T-cell therapies targeting CD19 if you have large B-cell lymphoma, follicular lymphoma, or mantle cell lymphoma. You may choose to receive other investigational therapy, if available. You may choose not to have treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

These alternative treatments have risks and benefits that may be the same or different than those in this research study. The study doctor can discuss these alternative treatments, including their risks and benefits with you.



The following is more detailed information about this study in addition to the information listed above.

#### Who can I talk to if I have questions or concerns?

If you have questions, concerns, or complaints, or think the research has hurt you, talk to the study doctor, Dr. Sattva Neelapu, at 713-792-2860.

This research has been reviewed and approved by an Institutional Review Board (IRB – an ethics committee that reviews research studies). You may talk to them at (713) 792-6477 or IRB Help@mdanderson.org if:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You want to talk to someone besides the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

#### How many people will be in this study?

It is expected about 33 people will be enrolled in this study. All will be enrolled at MD Anderson.

#### What happens if I agree to be in this research?

#### **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible.

- You will have a physical exam.
- You will have a neurological exam (tests to check the functioning of your nerves, including tests of your balance and reflexes).
- You will have an EKG and an echocardiogram (ECHO) to check your heart function.
- Blood (up to 3 tablespoons) will be drawn for routine tests and tests to check for HIV and hepatitis. If you have previously received treatment with CD19 CAR Tcell therapy, part of this sample will be used to check for CD19 CAR T-cell levels in your blood.
- You will have imaging scans with contrast (such as PET/CT, CT scans, or MRI, depending on what the doctor thinks is needed) to check the status of the disease.
- You will have a tumor biopsy to check the status of the disease. The study doctor will tell you the type of biopsy you will have.
- If the doctor thinks it is needed, you may have a bone marrow biopsy/aspirate to check the status of the disease. To collect a bone marrow biopsy/aspirate, an



- area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.
- If you can become pregnant, part of the above blood sample or a urine sample will be collected for a pregnancy test. To take part in this study, you must not be pregnant.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in the study, you will not be enrolled. Other options will be discussed with you.

#### **Study Groups**

There are 2 parts to this study: Part 1 (dose escalation) and Part 2 (dose expansion). If you are found to be eligible to take part in this study, you will be assigned to either Part 1 or Part 2 depending on when you join the study.

If you are enrolled in Part 1, the dose of JV-213 you receive will depend on when you join this study. Up to 3 dose levels of JV-213 will be tested. About 3-6 participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level of JV-213. Each new group will receive a higher dose of JV-213 than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of JV-213 is found.

If you are enrolled in Part 2, you will receive JV-213 at the recommended dose that was found in Part 1.

The study doctor will know what dose of JV-213 you are receiving, but neither you nor your doctor can decide which dose you will receive.

#### Leukapheresis

You will return to the clinic to have a **leukapheresis procedure** performed in order to collect enough white blood cells (T cells) to make the study product. For this procedure, you will need to stay seated in a chair and keep both arms still for about 3 hours. During this process, your blood will flow into the machine and then directly back into your bloodstream through the second line. Blood will be drawn from 1 arm through a catheter (needle and tube) connected to the leukapheresis machine. Inside the machine, the white blood cells (T cells) will be separated from the rest of the blood cells and collected in a sterile bag. Then, the rest of the blood cells will be returned through a catheter to your other arm. A blood thinner called citrate will be added to the blood as it enters the machine in order to lower the risk of your blood clotting in the machine.

The T cells that are collected will then be sent to a manufacturing facility to be genetically modified in order to make JV-213.

After the JV-213 is made, it is sent back to your study doctor so you may receive it.

At this visit, blood (about 1 tablespoon) will also be drawn for routine testing.



- Negative (or minus) days are days before you receive JV-213.
  - Day 0 is the day you receive JV-213.
  - Positive days are the days after you receive JV-213.

#### **Bridging Therapy (optional)**

If the doctor thinks it is needed, you may receive bridging therapy with chemotherapy, radiation therapy, biologic therapy, or corticosteroids for the disease before the start of conditioning therapy. If bridging therapy is given to you, the study doctor will explain how the drugs are given and their risks. Then, after you complete bridging therapy:

- You will have a PET-CT scan to check the status of the disease.
- Blood (up to 2 tablespoons) will be drawn to confirm you are still eligible to take part in the study.

#### Conditioning Therapy

On **Day -5 through Day -3**, you will receive conditioning chemotherapy (fludarabine and cyclophosphamide). This type of chemotherapy is given to help prepare your body and immune system to receive JV-213 cells. It is not meant to treat the cancer. You will receive fludarabine by vein over about 30 minutes for 3 days. You will also receive cyclophosphamide by vein over about 1 hour for about 3 days.

#### JV-213

You will receive JV-213 by vein over about 1 hour (or less) on **Day 0**. You may be hospitalized for at least 7 days while you are receiving JV-213 so the study team can watch you for side effects. If the study doctor thinks it is needed, you may stay in the hospital for a longer period.

After you leave the hospital, you will need to stay close to MD Anderson until about Day 28 after your JV-213 infusion.

If needed, you will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

#### Study Visits

**If, at any time during the study**, the doctor thinks it is important for your health, you may have an unscheduled visit. At this visit, some or all of the below tests/procedures may be done. This will be discussed with you.

In this study, blood will be drawn for routine and research tests. "Research tests" refers to the following:

- To check the status of the disease and how the drug is affecting the disease,
- Biomarker testing—Biomarkers are found in the blood/tissue and may be related to your reaction to the study drug. In this study, biomarker testing will also help researchers measure how much study drug is in the body at different time points



- To learn more about how your immune system and the study drug works together, and
- To learn more about how your genetic information (DNA) affects your response to the study drug(s).

On **Day -5**, or up to 72 hours before you receive conditioning chemotherapy:

- You will have a physical exam.
- Blood (up to 3 tablespoons) will be drawn for routine and research tests.
- If you can become pregnant, urine or part of the above blood sample will be collected for a pregnancy test.

On **Day 0** (the day you receive the CAR T cells):

- You will have a physical exam, including a neurological exam.
- Blood (up to 2 tablespoons) will be drawn for routine and research tests.

On Days 1-7, every other day during Days 8-14, and then on Days 21 and 28, you will have some or all of the following tests/procedures to check on your health:

- You will have a physical exam, including a neurological exam.
- Blood (up to 2 tablespoons per visit) will be drawn for routine and research tests.
- Between Days 7 and 14, you will have a tumor biopsy for research tests.
- On Day 28 only:
  - You will have a bone marrow biopsy if your screening bone marrow was positive for lymphoma and PET-CT scan does not show any evidence of lymphoma. (Day 28 only).
  - You will have a PET-CT imaging scan to check the status of the disease.

#### Follow-Up Visits and End-of-Study Visit

At **Month 2** after your dose of JV-213 you will have a follow-up visit for physical exam and routine blood test (1 tablespoon).

At **Months 3, 6, 9, 12, 18, and 24** after your dose of JV-213 you will have follow-up visits. At each visit:

- You will have a physical exam. At Month 3, you will also have a neurological exam
- Blood (up to 2 tablespoons per visit) will be drawn for routine and research tests.
- You will have imaging scans (such as an MRI, CT, or PET/CT depending on what the doctor thinks is needed) to check the status of the disease.
- You will have a bone marrow biopsy if your screening bone marrow was positive for lymphoma and PET-CT scan does not show any evidence of lymphoma.
- If the disease comes back or if the tumor increases in size after receiving JV-213, you may have a tumor biopsy for research tests.

**If you leave the study early**, you will come to the clinic within 14 days after your decision to leave the study to have the above tests/procedures.



To take part in this study, you must agree to participate in long-term follow-up, which will last about 15 years. During long-term follow-up beyond year 2, you will come to the clinic 1 time every year for the below tests/procedures. After Year 5, follow-up may be done as an in-person clinic visit or by video/telephone encounter or by mailed questionnaire. If by video/telephone, each call should last about 10-15 minutes.

#### At each follow-up visit:

- You will have a physical exam.
- Blood (up to 2 tablespoons per visit) may be drawn for routine and research tests.

#### What are my responsibilities if I take part in this research?

If you take part in this research, you will be responsible for the following:

- Tell the study doctor/study staff about all medications that you are taking or plan to take, including prescription and over-the-counter medications, supplements, vitamins, and herbal remedies.
- If you cannot attend an appointment, please contact the study team as soon as possible to schedule a new appointment.
- Tell the study staff about any symptoms, changes in medications, doctor's or nurse's appointments, or hospital admissions that you may have had.
- Do NOT participate in any other research study while you are in this study.
- Tell your primary doctor that you are taking part in this study.

#### What happens if I say yes, but I change my mind later?

You can leave the research at any time; it will not be held against you.

You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can then decide if you need to have any visits or tests to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can collect data from your routine medical care. If you agree, this data will be handled the same as research data.

## Is there any way being in this study could be bad for me? (Detailed Risks)

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are



rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

Conditioning chemotherapy and JV-213 may cause low blood cell counts (red blood cells, platelets, and white blood cells):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue.
   You may need a blood transfusion.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). You may need a platelet transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become lifethreatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing.

It is possible the study team may not be able to manufacture the JV-213 product. In such a situation, you will not be able to receive JV-213 treatment. It is also possible that sometimes the JV-213 cell dose manufactured is lower than the target dose. If this happens, your doctor will discuss with you whether it is appropriate to move forward with treatment with a lower cell dose of JV-213 but you will have the option to agree to move forward or decline and choose alternative treatment option outside of this study.

#### JV-213 Side Effects

This is the first study of JV-213 in humans, so the side effects are not well known.

Based on similar cell therapies, JV-213 may cause cytokine release syndrome (CRS). This involves a release of a large amount of proteins into the blood stream. This may cause changes in blood pressure and heartbeat, flu-like symptoms (nausea, fever, and chills), and/or affect your lung/liver/kidney function. It may also cause certain brain-related symptoms, such as dizziness, weakness, confusion, difficulty speaking, and/or decreased brain function (possible paralysis and/or coma).

Other side effects may include:

| <ul><li>confusion</li><li>difficulty</li><li>communicating,</li></ul> | <ul><li>low blood cell count<br/>(red, white, platelet)</li><li>allergic reaction</li></ul> | Tumor Lysis Syndrome (TLS) breakdown products |
|---|---|---|
| learning, and/or | (possible difficulty | of the cancer cells |
| comprehending | | entering the blood |
| speech | | stream (possible |



- loss of alertness
- headache
- anxiety
- difficulty sleeping
- dizziness
- muscle weakness
- tremors
- seizures
- brain swelling (possible headache and/or mental status changes)

- breathing, skin rash, fever, muscle/join pain, swelling)
- infusion reaction (fever, chills, and/or low blood pressure)
- immune system reaction (possible fever, jaundice, liver/spleen enlargement, irritability, and/or seizures)
- weakness, low blood pressure, muscle cramps, kidney damage, and/or other organ damage)
- infection

JV-213 may cause hemophagocytic lymphohistiocytosis/macrophage activation syndrome (HLH/MAS), which is an immune system reaction (possible fever, jaundice, liver/spleen enlargement, irritability, and/or seizures) that often results in death.

JV-213 is produced by using a virus called a lentivirus to genetically change the white blood cells collected by leukapheresis. The lentivirus is also changed to prevent it from multiplying and infecting your body after the JV-213 T cell product is given back to you. However, it is technically possible that it could cause an infection.

The act of genetically changing cells to produce JV-213 could cause genes to be transferred to cells where they could cause harm. This could cause you to develop another type of cancer (such as leukemia, a type of blood cancer).

#### **Conditioning Chemotherapy Side Effects**

The most common side effect of conditioning chemotherapy is a low blood cell count (red, platelets, and/or white blood cells). It may also cause abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure). Stroke (which may be fatal) has also been reported.

#### Commonly (in more than 20% of patients), cyclophosphamide may cause:

- headache
- hair loss (partial or total)
- mouth blisters/sores (possible difficulty swallowing)
- nausea/vomiting
- inability to regulate water/salt balance which can cause frequent urination and dehydration
- abdominal pain

- loss of appetite
- diarrhea
- problems with production of sperm and eggs
- inability to have children
- stopped menstrual cycle
- low blood counts (red, platelet, white)
- fever with dangerously low white blood cell count (febrile neutropenia)
- bladder inflammation and bleeding (possible pain and/or urge to urinate)
- infection



Cyclophosphamide may cause you to develop another type of cancer (such as bladder cancer, acute leukemia [a type of blood cancer], lymphoma [a type of lymph node cancer], thyroid cancer, and/or sarcoma [a type of cancer that can start in the soft tissue, bone, or other tissue].

### Rare but serious (occurring in fewer than 3% of patients), cyclophosphamide may cause:

- irregular heartbeat
- build-up of fluid around the heart (possible heart failure)
- build-up of blood in the sac around the heart (possible impaired heart function)
- inflammation of the heart and/or the tissue around the heart (possible chest pain and/or bleeding)
- heart damage/failure, death of heart tissue, or other severe heart problems
- heart attack, which can be serious and lifethreatening
- blood clots in a vein (possible pain, swelling, and/or redness)
- blood clots in an artery (possible organ damage such as stroke and/or heart attack)
- brain injury that may be reversible (possible headache, confusion, seizures, and/or vision loss)
- dizziness
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- severe sunburn-like rash at site of previous

- wound healing problems
- low blood levels of potassium (possible weakness)
- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)
- hormonal deficiency that affects the body's ability to control blood pressure and react to stress
- decreased supply of blood to the abdomen
- digestive system bleeding
- enlarged bowel (possible abdominal pain)
- inflammation of the intestines (possible bleeding)
- inflammation of the pancreas (possible abdominal pain)
- liver damage (possibly due to blood clots)
- jaundice (yellowing of skin and/or eyes)
- high blood levels of uric acid (possible painful joints and/or kidney failure)
- ovarian scarring
- urinary tract or bladder scarring

- hearing loss
- breakdown of muscle tissue (possible kidney failure)
- death of kidney tissue (possible kidney failure)
- difficulty breathing
- lung inflammation (possible difficulty breathing)
- problems with blood carrying oxygen (possible blue skin)
- lung damage due to blood clots
- increased blood pressure in the lungs (possible difficulty breathing and/or heart failure)
- multiorgan failure
- breakdown products of the cancer cells entering the blood stream (possible weakness, low blood pressure, muscle cramps, kidney damage, and/or other organ damage)
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)
- severe life-threatening infection (possible low



| radiation (called radiation recall) • very severe blistering skin disease (loss of large portion of skin) | <ul> <li>decreased testicle size and function</li> <li>blood in the urine</li> <li>blurry vision</li> </ul> | blood pressure, kidney<br>failure, and/or heart<br>failure) |
|---|---|---|
|---|---|---|

#### Commonly (in more than 20% of patients), fludarabine may cause:

| • fever | <ul><li>nausea</li></ul> | <ul><li>weakness</li></ul> |
|---|---|---|
| fatigue | <ul><li>vomiting</li></ul> | difficulty breathing |
| • pain | <ul> <li>low blood cell count</li> </ul> | • cough |
| <ul> <li>loss of appetite</li> </ul> | (red, white, platelets) | <ul><li>infection</li></ul> |

#### Occasional (occurring in 3-20% of patients), fludarabine may cause:

| <ul> <li>chest pain (possibly due to heart trouble)</li> <li>heart failure</li> <li>heart attack</li> <li>fast and/or irregular heartbeat</li> <li>blood clots in a vein (possible pain, swelling, and/or redness)</li> <li>vein inflammation</li> <li>swelling</li> <li>chills</li> <li>skin rash and/or itching</li> <li>sweating</li> <li>hair loss (partial or total)</li> <li>high blood sugar (possible diabetes)</li> <li>mouth blisters/sores (possible difficulty swallowing)</li> <li>diarrhea/constipation</li> <li>digestive system bleeding</li> <li>difficulty sleeping</li> <li>skin rash and/or itching</li> <li>sweating</li> <li>hair loss (partial or total)</li> <li>abnormal liver tests (possible liver damage)</li> <li>abnormal sensation (such as pins and needles)</li> <li>vision problems</li> <li>hearing loss</li> <li>sore/swollen throat</li> <li>lung damage/inflammation (possible difficulty breathing)</li> <li>coughing up blood</li> </ul> | | | | |
|---|---|---|---|---|
| | • | heart trouble) heart failure heart attack fast and/or irregular heartbeat blood clots in a vein (possible pain, swelling, and/or redness) vein inflammation swelling chills stroke headache | <ul> <li>itching</li> <li>sweating</li> <li>hair loss (partial or total)</li> <li>high blood sugar (possible diabetes)</li> <li>mouth blisters/sores (possible difficulty swallowing)</li> <li>diarrhea/constipation</li> <li>digestive system bleeding</li> <li>gallstones</li> <li>blood in the urine</li> </ul> | <ul> <li>abnormal liver tests (possible liver damage)</li> <li>abnormal sensation (such as pins and needles)</li> <li>vision problems</li> <li>hearing loss</li> <li>sore/swollen throat</li> <li>lung damage/inflammation (possible difficulty breathing)</li> </ul> |

#### Rare but serious (occurring in fewer than 3% of patients), fludarabine may cause:



- abnormal brain function (affecting balance and coordination)
- progressive multifocal leukoencephalopathy (PML – a disease with brain damage that may likely result in paralysis and/or coma, which may be permanent, or death)
- mental status change
- coma
- seizure
- abnormal salts, minerals, and/or acid levels in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)

- bladder inflammation with bleeding (possible pain and/or urge to urinate)
- bone marrow failure due to abnormal tissue growth
- destruction of red blood cells and platelets due to abnormal antibodies
- anemia due to destruction of red blood cells
- condition causing increased bleeding and/or bruising
- liver failure
- nerve damage (possible numbness, pain, and/or loss of motor function)

- painful joints and/or kidney failure)
- bleeding in the lungs and/or airways
- failure to breathe
- low oxygen level in the blood (possible lightheadedness)
- life-threatening allergic reaction (such as difficulty breathing, low blood pressure, and/or organ failure)
- breakdown products of the cancer cells entering the blood stream (possible weakness, low blood pressure, muscle cramps, kidney damage, and/or other organ damage)

Fludarabine may rarely cause you to develop another type of cancer (such as skin cancer and/or acute myeloid leukemia [a type of blood cancer].

The study doctor can discuss the other risks of conditioning chemotherapy.

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

#### Other Side Effects

#### **Leukapheresis Side Effects**

It is not well known how often the following side effects may occur.



- low blood pressure (possible dizziness/fainting)
- chest discomfort
- irregular heartbeat
- heart failure
- chills
- shock
- seizure
- fainting
- anxiety
- fatigue

- tingling and/or numbness
- dizziness
- low blood levels of calcium (possible weakness and/or cramping)
- nausea
- vomiting
- low blood counts (red, platelets)
- destruction of red blood cells

- difficulty breathing
- air entering the blood stream
- loss of blood (if the tubing breaks or the machine malfunctions)
- discomfort, bruising, bleeding, and/or infection at the needle insertion site
- infection

Citrate may cause numbness and/or tingling of the fingertips and/or around the mouth, weakness, and/or severe muscle cramps. Tell the study staff right away if you have any numbness/tingling, weakness, chills, and/or stiff arms.

You should avoid all aspirin and ibuprofen products for at least 3 days before and also during the leukapheresis procedures. Any high physical activity, especially contact sports such as football and basketball, should be avoided for 24 hours after the leukapheresis procedure.

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **bone marrow biopsies/aspirates and tumor biopsies** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**EKGs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

All drugs have a potential risk of causing an **allergic reaction**, which (if not treated quickly) could become life-threatening. You should get medical help and contact the study doctor right away if you think you have any of the following symptoms of a serious allergic reaction:

- trouble breathing or
- swelling of the face, mouth, lips, gums, tongue, or neck.
- Other allergic reactions may include rash, hives, or blisters.

During an **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or



closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

A **PET/CT** scan may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort or the scanning will be stopped.

The PET/CT scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

Although every effort will be made to keep **study data** safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets during the study and will continue to be stored securely after the study. Only authorized people who are working on this study will have access to study data.

This research project may impact your fitness for duty. Please seek command or Component guidance before participating.

This research includes the potential risk of the loss of clearance, credentials, or other privileged access or duty.



In addition to these risks, this research may hurt you in ways that are unknown. These may be a minor inconvenience or may be so severe as to cause death.

You will be told about any new information that may affect your health, welfare, or choice to stay in the research.

#### **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child after you are enrolled on this study and for at least 6 months after JV-213 therapy.

If you can become pregnant or father a child, you must use birth control starting at least 1 month before conditioning chemotherapy and then through at least 6 months after JV-213 therapy, if you are sexually active.

If you are male and your partner can become pregnant or is currently pregnant or breastfeeding, even if you have undergone a successful vasectomy, you must agree to use a condom and your partner must also use at least 1 method of birth control.

If you can become pregnant, you must use 2 reliable forms of birth control (1 highly effective method and 1 additional effective method at the same time).

# Highly Effective Methods Intrauterine Device (IUD) Hormonal (birth control pills, injections, implants) Bilateral tubal occlusion/ligation (also known as having your "tubes tied") Partner's vasectomy

## Additional Effective Methods Latex Condom Diaphragm Cervical cap

Birth control methods are not perfect, even when used properly. If you or your partner become pregnant during the study, or you want to stop your required birth control during the study, you should tell the study doctor right away.

**Males**: Do not donate sperm during the study and for at least 6 months after JV-213 therapy. Tell the doctor right away if your partner becomes pregnant or suspects pregnancy. If your partner/spouse becomes pregnant while you are on this study, the sponsor would like to collect information about the pregnancy. The study sponsor's contact information will be made available so that, if you and your partner wish to, you can share information about the outcome of the pregnancy with the sponsor. If you and/or your partner choose not to share this information, it will not result in any penalty or loss of benefits to which you are otherwise entitled.



**Females**: If you are pregnant, you will not be enrolled on this study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away. The sponsor will ask for information about the pregnancy.

If you become pregnant, no additional anti-cancer therapy will be administered on the study, but you will be monitored for long-term follow-up as part of this study.

## Will it cost anything to be in this study? Will I be paid to be in this study?

JV-213 will be provided at no cost to you during the study. You and/or your insurance provider will be responsible for the cost of conditioning chemotherapy (cyclophosphamide and fludarabine) and for any hospitalizations.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

You will not receive any compensation for taking part in this study.

#### What happens to the information collected for the research?

Efforts will be made to limit the use and disclosure of your personal information, including research study and medical records, to people who need to review this information. Complete secrecy cannot be promised. Organizations that may inspect and copy your information include the IRB and other representatives of this organization.

A participant study number will be assigned to you once you have been enrolled in the study. This participant study number will be used to identify your data in the study report and when reporting any data from the study.

Any personal information that could identify you will be removed or changed before data are shared with other researchers or results are made public.

The study is partly supported by the Department of Defense Medical Research Program. The sponsor, monitors, auditors, the IRB, Department of Defense, and the Food and Drug Administration will be granted direct access to your medical records to conduct and oversee the research. By signing this document, you are authorizing this



access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

Federal law provides additional protections of your medical records and related health information. These are described below.

#### Will my data or samples be used for future research?

Your personal information and/or samples are being collected as part of this study. These data and/or samples may be used by researchers at MD Anderson or shared with other researchers and/or institutions for use in future research.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the MD Anderson IRB before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

If identifiers are removed from your identifiable private information or identifiable samples that are collected during this research, that information or those samples could be used for future research studies or shared with another researcher for future research studies without your additional informed consent.

#### Can I be removed from the research study without my permission?

The person in charge of the research study can remove you from the research study without your approval. Possible reasons for removal include if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

#### What happens if I get hurt from being in this study?

If you get sick or hurt and it is related to your participation in this study, you will be given care at MD Anderson (if you are at the clinic when you are sick or hurt). If you get hurt or sick and you are not at the clinic (for example, you are at home or at another doctor's office):

- call your personal doctor right away (or in an emergency, call 911)
- tell your personal doctor or ER staff that you are in this study (try to give them a copy of this consent form or show them your participant card)
- call the study doctor (Dr. Sattva Neelapu, at 713-792-2860)

You will not be reimbursed for expenses or compensated financially by MD Anderson for this injury. Costs of treatment received because you were hurt or sick will be billed to you or your insurance company. No other form of payment is available.



You may also contact the MD Anderson IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

#### What else do I need to know?

MD Anderson may benefit from your participation and/or what is learned in this study.

Your information and samples (both identifiable and de-identified) may be used to create products or to deliver services, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will contact you to let you know what they have found. If the researchers return genetic test results to you, it may be because they think you could have a health risk and want to recommend that the test should be re-done by a certified clinical laboratory to check the results. If this happens, then you may want to get a second test from a certified clinical laboratory, consult your own doctor, or get professional genetic counseling. You may have to pay for those additional services yourself.

This research study involves genetic testing. The Genetic Information Nondiscrimination Act (GINA) prohibits health insurers or health plan administrators from requesting or requiring genetic information of you or your family members, or using such information for decisions regarding your eligibility for insurance or your premiums. However, this law does <u>not</u> provide the same protection for disability, life insurance, or long-term care insurance. GINA also prohibits most employers (with 15 employees or more) from using genetic information when making decisions on your employment, including decisions related to hiring, firing, promotion, pay, and job assignments. Please contact the study doctor if you would like more information about GINA and how it protects you from genetic discrimination.

#### **Optional Procedures for the Study**

You do not have to agree to the optional procedure(s) in order to take part in this study. There are no benefits to you for taking part in the optional procedures. Future patients may benefit from what is learned. You may stop taking part at any time. There will be no cost to you for taking part in the optional procedures.

**Optional Procedure #1:** If you agree, you will have a tumor biopsy about 7-14 days after JV-213 infusion. The tissue will be used to help researchers understand how JV-213 is affecting the disease. The tissue may be stored by MD Anderson for about 15 years. At any time, you may contact your study doctor in writing and request that the samples be destroyed. If you decide to stop participating in the study, but do not request



that your samples be destroyed, the sponsor may continue to use your samples for research as described above.

**Optional Procedure #2:** If you agree, leftover blood and tissue samples will be stored by MD Anderson Cancer Center and/or Cell Therapy Manufacturing Center for up to 15 years for future research related to the treatment or the disease. If you later change your mind about use of these samples for future research, tell the study doctor in writing that you want the samples destroyed.

**Optional Procedure Risks:** Having a **tumor biopsy** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

The use of **leftover blood and tissue samples for future research** is not expected to cause any additional risks for you.

CONSENT/PERMISSION/AUTHORIZATION FOR OPTIONAL PROCEDURES Circle your choice of "yes" or "no" for each of the following optional procedures:

**Optional Procedure #1:** Do you agree to have a tumor biopsy to help researchers understand how the study drug affects the disease?

YES NO

**Optional Procedure #2:** Do you agree to have leftover blood and tissue samples to be used for future research related to the treatment or the disease?

YES NO

## Authorization for Use and Disclosure of Protected Health Information (PHI):

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], Department of Defense, and OHRP)
  - The IRB and officials of MD Anderson
  - Cell Therapy Manufacturing Center (CTMC)
  - Any future sponsors/supporters of the study, and/or licensees of the study technology
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form



The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.
  - Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.



#### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document.

| SIGNATURE OF PARTICIPANT | DATE |
|---|---|
| | _, _, |
| PRINTED NAME OF PARTICIPANT | |
| WITNESS TO CONSENT I was present during the explanation of the research to be performed | I under this protocol. |
| SIGNATURE OF WITNESS TO THE VERBAL CONSENT PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. | DATE |
| PRINTED NAME OF WITNESS TO THE VERBAL CONSENT | |
| PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or representative, using language that is understandable and appropriate have fully informed this participant of the nature of this study and its and risks and that the participant understood this explanation. | te. I believe that I |
| PERSON OBTAINING CONSENT | DATE |
| PRINTED NAME OF PERSON OBTAINING CONSENT | |